CLINICAL TRIAL: NCT02618733
Title: A Prospective Randomized Controlled Clinical Trial of Comparing ticagreLor Versus clopidogrEl on mIcrocirculation in Patients With Acute cOronary Syndrome Study
Brief Title: Comparing Ticagrelor Versus Clopidogrel on Microcirculation
Acronym: PLEIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dong-A University (Other)
Collaborators: AstraZeneca (Industry); Biotronik SE & Co. KG (Industry)
Responsible Party: Principal Investigator, Kyungil Park, Assistant professor, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-218
Record Dates: First submitted 2015-11-25; First posted 2015-12-01 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 90mg, twice a day
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Clopidogrel 75mg, once a day
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — 90mg, twice a day
  Arms: Ticagrelor
Drug: Clopidogrel — 75mg, once a day
  Arms: Clopidogrel

SUMMARY:
Recently, data (PLATO) from an AstraZeneca study of platelet inhibition and patient outcomes, a Phase III pivotal efficacy and safety study with a duration of up to 12 months comparing ticagrelor 90 mg twice daily dosing to clopidogrel 75 mg once daily dosing in acute coronary syndrome patients on ASA background, have demonstrated superiority of ticagrelor over clopidogrel in the prevention of fatal and non-fatal cardiovascular events. Currently, the mechanism for this mortality reduction remain uncertain. One hypothesis is a adenosine mediated theory that ticagrelor has been shown to enhance adenosine-induced vasodilation. Several experimental and clinical studies support the hypothesis that adenosine could reduce cardiac ischaemia reperfusion damage. Moreover, recent study has demonstrated that ticagrelor enhances adenosine-induced coronary vasodilatory responses in healthy humans. However, there are no available data on coronary circulation effects after chronic treatment of ticagrelor in patients with ACS who have altered resting coronary blood flow dynamics due to advanced coronary artery disease.

DETAILED DESCRIPTION:
This study is a prospective, randomized, open-label, active controlled study with two parallel study groups.

For inclusion in the study subjects should fulfill the following criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female or male aged 20-85 years
3. All patients with ACS scheduled for PCI will be eligible, assuming their ability to understand the character and individual consequences of participation as well as giving written informed consent.
4. Be able to understand and comply with the requirements of the study, as judged by the investigator.

To investigate the effects of ticagrelor on coronary microcirculation, IMR will be measured twice, 6 months apart in the same lesion, compared with clopidogrel.

The IMR is defined as simultaneously measured distal coronary pressure divided by the inverse of the thermodilution-derived hyperaemic mean transit time (Tmn), or more simply, distal coronary pressure multiplied by the Tmn.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* All patients with ACS scheduled for PCI will be eligible, assuming their ability to understand the character and individual consequences of participation as well as giving written informed consent.
* Be able to understand and comply with the requirements of the study, as judged by the investigator.

Exclusion Criteria:

* History of intracranial bleeding
* Severe hepatic impairment
* Active pathologic bleeding
* Hypersensitivity to ticagrelor or any of the excipients
* Liver cirrhosis greater than or equal to Child class B
* Decreased serum platelet level (≤ 100,000/uL)
* Life expectancy ≤ 1 year
* Need for chronic oral anticoagulant therapy
* Patients with known bleeding diathesis or coagulation disorder
* History of previous intracranial bleed at any time, gastrointestinal bleed within the past 6 months, or major surgery within 30 days.
* Ischemic stroke within the previous 14 days
* Renal failure requiring dialysis or anticipated need for dialysis during the course of the study
* Concern for inability of the patient to comply with study procedures and/or follow up
* Unable to give informed consent.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Index of microcirculatory resistance using 0.014-in coronary pressure wire | 6 months

SECONDARY OUTCOMES:
Fractional flow reserve using 0.014-in coronary pressure wire | 6 months
Coronary flow reserve using 0.014-in coronary pressure wire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kyungil Park, MD, Study Director — Dong-A University
Locations (1):
- Department of Internal Medicine,Dong-A University College of Medicine, Busan, South Korea

REFERENCES:
- [Derived] Moon H, Jo YS, Kim SJ, Jo S, Park K. Comparison of ticagrelor with clopidogrel on quality of life in patients with acute coronary syndrome. Health Qual Life Outcomes. 2021 Oct 16;19(1):242. doi: 10.1186/s12955-021-01875-w. PMID 34656119
- [Derived] Jeong YJ, Park K, Kim YD. Comparison between ticagrelor and clopidogrel on myocardial blood flow in patients with acute coronary syndrome, using 13 N-ammonia positron emission tomography. Am Heart J. 2020 Apr;222:121-130. doi: 10.1016/j.ahj.2020.01.013. Epub 2020 Jan 27. PMID 32028138
- [Derived] Park K, Cho YR, Park JS, Park TH, Kim MH, Kim YD. Comparison of the Effects of Ticagrelor and Clopidogrel on Microvascular Dysfunction in Patients With Acute Coronary Syndrome Using Invasive Physiologic Indices. Circ Cardiovasc Interv. 2019 Oct;12(10):e008105. doi: 10.1161/CIRCINTERVENTIONS.119.008105. Epub 2019 Sep 26. PMID 31554423